CLINICAL TRIAL: NCT00678418
Title: Efficacy and Safety of VIVITROL® (Naltrexone for Extended-release Injectable Suspension) in Adults With Opioid Dependence
Brief Title: ALK21-013: Efficacy and Safety of Medisorb® Naltrexone (VIVITROL®) in Adults With Opioid Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK21-013
Record Dates: First submitted 2008-05-14; First posted 2008-05-15 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Opiate Dependence
Keywords: Addiction; Opiate dependence; Inpatient detoxification; opioid dependence; heroin dependence
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Heroin Dependence | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIVITROL® 380 mg (Experimental)
  Interventions: Drug: VIVITROL® 380 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIVITROL® 380 mg — Administered via intramuscular (IM) injection once every 4 weeks for 24 weeks during Part A, followed by once every 4 weeks for 52 weeks in Part B.
  Other Names: Naltrexone for extended-release injectable suspension; Medisorb® naltrexone
  Arms: VIVITROL® 380 mg
Drug: Placebo — Administered via IM injection once every 4 weeks for 24 weeks during Part A, followed by VIVITROL® 380 mg via IM injection once every 4 weeks for 52 weeks in Part B.
  Arms: Placebo

SUMMARY:
This is a Phase 3 multi-center trial designed to evaluate the clinical efficacy and safety of VIVITROL® (Medisorb® naltrexone 380 mg) versus placebo when administered to adults upon discharge from inpatient treatment for opioid dependence.

The study was conducted in 2 parts, Part A and Part B. The clinical portion of both parts has completed. Results for Part B are not yet available.

DETAILED DESCRIPTION:
Part A was a double-blind, randomized, placebo-controlled assessment of the efficacy and safety of 24 weeks of monthly treatment with VIVITROL compared to placebo in opioid-dependent adults.

Subjects who completed Part A could choose to continue to Part B, which was an open-label extension to assess longer-term safety, durability of effect, health economics, and quality of life (QOL) in the continuing study population for up to 1 year.

At the conclusion of both parts, each completing subject will have received a total of up to 19 injections of study drug over approximately 1.5 years.

Dosing was performed by the principal investigator or designated study staff member.

All subjects received standardized, manual-based psychosocial support at each scheduled visit. Opioid use was tracked through urine drug testing and subjects' self reports. Other evaluations for efficacy and safety, health economics, and quality of life were routinely conducted throughout the study.

ELIGIBILITY:
Primary Inclusion Criteria:

* Written, informed consent
* 18 years of age or older
* Current diagnosis of opioid dependence, based on Diagnostic and Statistical Manual of Mental Health Disorders, 4th Ed. (DSM-IV-TR) criteria
* Voluntarily seeking treatment for opioid dependence
* Completing or recently completed up to 30 days of inpatient treatment for opioid detoxification, and off all opioids (including buprenorphine and methadone) for at least 7 days
* Noncustodial, stable residence and phone, plus 1 contact with verifiable address and phone
* Significant other (eg, spouse, relative) willing to supervise compliance with the study visit schedule and procedures
* Agree to use contraception for study duration if of childbearing potential

Primary Exclusion Criteria:

* Pregnancy or lactation
* Clinically significant medical condition or observed abnormalities (eg: physical exam, electrocardiogram (ECG), lab and/or urinalysis findings)
* Positive naloxone challenge test at randomization (Day 0)
* Evidence of hepatic failure including: ascites, bilirubin >10% above upper limit of normal (ULN) and/or esophageal variceal disease
* Past or present history of an acquired immunodeficiency syndrome (AIDS)-indicator disease in HIV-infected subjects
* Active hepatitis and/or aspartate aminotransferase (AST), alanine aminotransferase(ALT) >3xULN
* Current major depression with suicidal ideation, psychosis, bipolar disorder, or any psychiatric disorder that would compromise ability to complete the study
* Recent history (within 6 months prior to screening) of suicidal ideation or attempt
* Dependence within prior year based on DSM-IV-TR, to any drugs other than prescription opioids or heroin, caffeine, marijuana, or nicotine
* Active alcohol dependence within prior 6 months
* Current alcohol use disorder that would, in the Investigator's opinion, preclude successful completion of the study
* Positive urine drug test for cocaine, benzodiazepines, or amphetamines at screening
* Use of oral naltrexone for 7 consecutive days within 60 days prior to screening
* Known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or polylactide-co-glycolide (PLG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Krupitsky, Prof., Principal Investigator — Leningrad Regional Addiction Center; Ruslan Ilyuk, Dr., Principal Investigator — Bekhterev Psychoneurological Research Institute; Edvin Zvartau, Prof., Principal Investigator — Saint-Petersburg State Medical University n.a. Pavlov; Alexander Sofronov, Prof., Principal Investigator — Saint-Petersburg Addiction Hospital; Alexey Egorov, Prof., Principal Investigator — Saint-Petersburg Addiction Hospital; Alexander Okhapkin, Prof., Principal Investigator — Addiction Treatment Center, Clinical Facility of Smolensk State Medical Academy; Nikolay Bokhan, Prof., Principal Investigator — Tomsk Mental Health Research Institute; Vladimir Mendelevich, Prof., Principal Investigator — Kazan State Medical University; Yuri Sivolap, Prof., Principal Investigator — Moscow Medical Academy n.a. I.M. Sechenov; Oleg Eryshev, Prof., Principal Investigator — Bekhterev Psychoneurological Research Institute; Nikolay Ivanets, Prof., Principal Investigator — National Addiction Scientific Center; Vitaliy Sinitskiy, Prof., Principal Investigator — Northern State Medical University; Andrey Anipchenko, Dr., Principal Investigator — Saint-Petersburg Addiction Hospital
Locations (1):
- Ethics Committee within the Federal Authority for Healthcare and Social Development Regulation, Moscow, Russia

REFERENCES:
- [Result] Krupitsky E, Nunes EV, Ling W, Gastfriend DR, Memisoglu A, Silverman BL. Injectable extended-release naltrexone (XR-NTX) for opioid dependence: long-term safety and effectiveness. Addiction. 2013 Sep;108(9):1628-37. doi: 10.1111/add.12208. Epub 2013 May 24. PMID 23701526
- [Result] Nunes EV, Krupitsky E, Ling W, Zummo J, Memisoglu A, Silverman BL, Gastfriend DR. Treating Opioid Dependence With Injectable Extended-Release Naltrexone (XR-NTX): Who Will Respond? J Addict Med. 2015 May-Jun;9(3):238-43. doi: 10.1097/ADM.0000000000000125. PMID 25901451
- [Result] Mitchell MC, Memisoglu A, Silverman BL. Hepatic safety of injectable extended-release naltrexone in patients with chronic hepatitis C and HIV infection. J Stud Alcohol Drugs. 2012 Nov;73(6):991-7. doi: 10.15288/jsad.2012.73.991. PMID 23036218
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Krupitsky E, Zvartau E, Blokhina E, Verbitskaya E, Wahlgren V, Tsoy-Podosenin M, Bushara N, Burakov A, Masalov D, Romanova T, Tyurina A, Palatkin V, Slavina T, Pecoraro A, Woody GE. Randomized trial of long-acting sustained-release naltrexone implant vs oral naltrexone or placebo for preventing relapse to opioid dependence. Arch Gen Psychiatry. 2012 Sep;69(9):973-81. doi: 10.1001/archgenpsychiatry.2012.1a. PMID 22945623
- [Derived] Krupitsky E, Nunes EV, Ling W, Illeperuma A, Gastfriend DR, Silverman BL. Injectable extended-release naltrexone for opioid dependence: a double-blind, placebo-controlled, multicentre randomised trial. Lancet. 2011 Apr 30;377(9776):1506-13. doi: 10.1016/S0140-6736(11)60358-9. PMID 21529928

RESULTS

PARTICIPANT FLOW:
Groups:
- VIVITROL® 380 mg; Placebo: Single intramuscular (IM) injection administered every 4 weeks
Period: Part A (Double Blind)
Arm/Group | VIVITROL® 380 mg | Placebo
Started | 126 | 124
Completed | 67 | 47
Not Completed | 59 | 77
Period: Part B (Open Label)
Arm/Group | VIVITROL® 380 mg | Placebo
Started | 114 (All participants who received placebo in Part A were switched to open-label VIVITROL in Part B.) | 0
Completed | 71 | 0
Not Completed | 43 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIVITROL® 380 mg | Placebo | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 124 | 250
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (4.8) | 29.7 (3.6) | 29.6 (4.2)
Gender [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 113 | 107 | 220
Region of Enrollment [Number; unit: participants]
  Russian Federation | 126 | 124 | 250

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Opioid-free Weeks Per Subject in Double-blind Period (Part A)
Description: Included are data from the last 20 weeks of the 24-week double-blind treatment period (Part A). Response profiles for each Arm are based on subjects' individual rates of weekly opioid-free data, including negative urine test results, attendance at study visits, and self-reports of opioid use/non-use.
Time Frame: 20 weeks
Population: Analyses include all randomized subjects who received at least 1 dose of study drug (Intent-to-treat [ITT] population).
Measure: Median (Inter-Quartile Range); unit: Percentage of opioid-free weeks
Arm/Group | VIVITROL® 380 mg | Placebo
Number analyzed (Participants) | 126 | 124
Percentage of opioid-free weeks | 90.0 (40.1) [20.0 to 100.0] | 35.0 (43.3) [0.0 to 95.0]
Statistical Analysis 1: Comparison: VIVITROL® 380 mg vs Placebo; Null hypothesis = the distribution function of opioid-free weeks is the same for both treatment groups; Test type: Superiority or Other; p = 0.0002, Van der Waerden

2. Secondary Outcome: Days to Discontinuation During Part A
Description: Defined as the duration of study participation and calculated as the number of days from Dose 1 to the day of study discontinuation.
Time Frame: 168 days (24 weeks)
Population: Analyses include all randomized subjects who received at least 1 dose of study drug (ITT population).
Measure: Median (95% Confidence Interval); unit: Days to study discontinuation
Arm/Group | VIVITROL® 380 mg | Placebo
Number analyzed (Participants) | 126 | 124
Days to study discontinuation | NA [NA to NA] — The median estimate for VIVITROL is >168 days (the duration of the treatment period). The median and confidence interval cannot be estimated because less than 50% of VIVITROL subjects discontinued during the 168-day treatment period. | 96.0 [63.0 to 165.0]
Statistical Analysis 1: Comparison: VIVITROL® 380 mg vs Placebo; P-value was calculated using the log-rank test for the null hypothesis: the distribution of days to discontinuation does not differ by treatment; Test type: Superiority or Other; p = 0.0042, Kaplan Meier — A total of 114 subjects continued on-study beyond the 168-day endpoint for Part A; these subjects were censored as of the first dosing day in Part B

3. Secondary Outcome: Craving Score: Change From Baseline
Description: Measured using subjects' response on a validated Visual Analog Scale at prespecified weekly visits throughout Part A, with comparison of baseline to end of Part A. The scale ranged from 0 ("No craving") to 100 ("highest possible craving").
Time Frame: Baseline to 6 months (24 weeks)
Population: Analyses include all randomized subjects who received at least 1 dose of study drug (ITT population).
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | VIVITROL® 380 mg | Placebo
Number analyzed (Participants) | 126 | 124
Units on a scale | -10.087 [-12.333 to -7.840] | 0.654 [-3.139 to 4.446]
Statistical Analysis 1: Comparison: VIVITROL® 380 mg vs Placebo; P-value was calculated using the Chi-square test for the null hypothesis: mean treatment difference = 0. Calculations were based on the Generalized Estimating Equation (GEE) model (normal distribution, identity link and AR(1) correlation structure) for repeated data on change from baseline with treatment and visit as main effects, and baseline as a covariate. Missing data were imputed using the Last Observation Carried Forward (LOCF) method; Test type: Superiority or Other; p < 0.0001, Chi-squared

4. Secondary Outcome: Incidence of Subjects Who Relapsed to Physiologic Opioid Dependence During the 24-week Treatment Period (Part A)
Description: Assessment of relapse to physiologic opioid dependence was based on individual subjects' results on the naloxone challenge test. A positive naloxone challenge test result was considered as a relapse to physiologic opioid dependence.
Time Frame: 24 Weeks
Population: Analyses include all randomized subjects who received at least 1 dose of study drug (ITT population).
Measure: Number; unit: Percentage of participants who relapsed
Arm/Group | VIVITROL® 380 mg | Placebo
Number analyzed (Participants) | 126 | 124
Percentage of participants who relapsed | 46.8 | 62.1
Statistical Analysis 1: Comparison: VIVITROL® 380 mg vs Placebo; Chi-square test was used to calculate the p-value for treatment. Null hypothesis = no association between relapse to dependence and study treatment. Subjects who discontinued prematurely from the study were imputed as having a positive naloxone challenge test result; Test type: Superiority or Other; p = 0.0154, Chi-squared; Risk Ratio (RR) = 0.75, 95% CI [0.60 to 0.95]

5. Secondary Outcome: Change in Percentage of Self-reported Opioid-free Days From Baseline to Week 24
Description: Opioid use was measured using subjects' entries on a validated Timeline FollowBack (TLFB) calendar in which they recorded their use/non-use of opioids each day.
Time Frame: 24 Weeks
Population: Analyses include all randomized subjects who received at least 1 dose of study drug (ITT population). Change from baseline was calculated per subject as the percent of subjects' self-reported opioid-free days in Part A minus the percent of opioid-free days prior to the subjects' hospitalization for pre-study detoxification.
Measure: Median (Inter-Quartile Range); unit: Percentage of opioid-free days
Arm/Group | VIVITROL® 380 mg | Placebo
Number analyzed (Participants) | 126 | 124
Percentage of opioid-free days | 75.83 [32.14 to 100.00] | 46.43 [11.01 to 96.76]
Statistical Analysis 1: Comparison: VIVITROL® 380 mg vs Placebo; Null hypothesis: Treatment difference=0. Missing data from subjects due to early discontinuation during Part A were imputed using the baseline rate; thus data for subjects who discontinued early were imputed as having no change from baseline; Test type: Superiority or Other; p = 0.0031, van der Waerden

ADVERSE EVENTS:
Time Frame: 6 Months (Part A)
Description: All participants who received at least 1 dose of randomized, double-blinded study drug (VIVITROL or placebo) are included in the safety population for Part A. Adverse events were tallied by number of participants affected as opposed to number of incidences reported for a given preferred term.
Arm/Group | VIVITROL® 380 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/126 | 4/124
Other Adverse Events (participants affected / at risk) | 63/126 | 40/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIVITROL® 380 mg (N=126) | Placebo (N=124)
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Adnexitis (Infections and infestations) | 1 | 0
HIV infection WHO clinical stage III (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIVITROL® 380 mg (N=126) | Placebo (N=124)
Alanine aminotransferase increased (Investigations) | 16 | 7
Aspartate aminotransferase increased (Investigations) | 13 | 3
Gamma-glutamyl transferase increased (Investigations) | 9 | 4
Nasopharyngitis (Infections and infestations) | 9 | 3
Influenza (Infections and infestations) | 6 | 5
Insomnia (Psychiatric disorders) | 8 | 1
Injection site pain (General disorders) | 6 | 1
Toothache (Gastrointestinal disorders) | 5 | 2
Hypertension (Gastrointestinal disorders) | 6 | 4
Headache (Nervous system disorders) | 4 | 3
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Drug dependence (Psychiatric disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 2
Transaminases increased (Investigations) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Pharyngolarnygeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Protein total increased (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual investigator may publish results until after the publication of the overall study without receiving Alkermes' written approval. After that time, a PI/Institution may publish results for noncommercial purposes. Should an investigator wish to do so, the Sponsor will have 30 days to review the proposed publication. The PI/Institution will delete any Sponsor Confidential Information other than study results and will revise a publication based on regulatory requirements of the Sponsor.